CLINICAL TRIAL: NCT01592136
Title: Expanded Access Program of Ponatinib (AP24534) for Patients With Refractory Chronic Myeloid Leukemia or Ph+ Acute Lymphoblastic Leukemia
Brief Title: Expanded Access Program of Ponatinib
Status: Approved for marketing | Type: Expanded Access
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: AP24534-12-901
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Chronic Myeloid Leukemia (CML); Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ ALL)
Keywords: Ponatinib; Tyrosine kinase inhibitor
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

INTERVENTIONS:
Drug: ponatinib — Patients will receive ponatinib 45 mg orally as a single dose once daily with or without food. Each patient will receive daily ponatinib until disease progression, unacceptable toxicity, or withdrawal of consent
  Other Names: AP24534

SUMMARY:
This protocol will allow expanded access of ponatinib to patients ≥18 years with chronic myeloid leukemia (CML) any phase or Philadelphia chromosome positive acute lymphoblastic leukemia (Ph+ALL) who have failed all available treatment options.

DETAILED DESCRIPTION:
This protocol will allow expanded access of ponatinib to patients ≥18 years with CML or Ph+ALL who have failed all available treatment options. Patients with chronic (CP) or accelerated phase (AP) CML must be previously treated with and resistant or intolerant to imatinib, dasatinib and nilotinib or develop the T315I mutation after any tyrosine kinase inhibitor (TKI) therapy. Patients with blast phase (BP) CML and Ph+ ALL must be previously treated with and resistant or intolerant to imatinib and dasatinib or develop the T315I mutation after any TKI therapy. No formal analysis will be performed on any data obtained. Safety information will be collected and adverse events will be tabulated for reporting purposes only.

ELIGIBILITY:
Main Inclusion Criteria:

1. CP-CML and AP-CML patients previously treated with and resistant or intolerant to imatinib, dasatinib and nilotinib or those who developed the T315I mutation after any TKI therapy. BP-CML and Ph+ ALL patients previously treated with and resistant or intolerant to imatinib and dasatinib or those who developed the T315I mutation after any TKI therapy.
2. Patients must be ≥ 18 years old.
3. Provide written informed consent.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Men and women of childbearing potential must agree to effective contraception from the time of signing informed consent through the Follow-up Visit, approximately 30 days after last dose of ponatinib.

Main Exclusion Criteria:

Patients are not eligible for participation in the study if they meet any of the following exclusion criteria:

1. Are eligible for an ongoing and accessible clinical trial of ponatinib
2. Have not adequately recovered from AEs due to agents previously administered
3. Require concurrent treatment with immunosuppressive agents, other than corticosteroids prescribed for a short course of therapy.
4. Have previously been treated with ponatinib.
5. Have significant or active cardiovascular disease, specifically including, but not restricted to:

   * Myocardial infarction within 3 months prior to first dose of ponatinib,
   * History of clinically significant atrial arrhythmia or any ventricular arrhythmia,
   * Unstable angina within 3 months prior to first dose of ponatinib,
   * Congestive heart failure within 3 months prior to first dose of ponatinib.
6. Have abnormal QTcF (> 450 ms for males or > 470 ms for females)
7. Have a significant bleeding disorder unrelated to CML or Ph+ ALL.
8. Have a history of pancreatitis or alcohol abuse
9. Have elevated amylase or lipase (> 1.5 x ULN for institution) at entry.
10. Have inadequate hepatic function or any of the following:

    * Total bilirubin > 1.5 x ULN for institution at entry
    * Alanine aminotransferase and aspartate aminotransferase > 2.5 x ULN for institution at entry
    * Prothrombin time >1.5 x ULN for institution at entry
11. Have inadequate renal function or serum creatinine > 2.5 x ULN for institution at entry
12. Have uncontrolled hypertriglyceridemia or triglycerides > 450 mg/dL at entry.
13. Have malabsorption syndrome or other gastrointestinal illness that could affect absorption of orally administered ponatinib.
14. Women who are pregnant or lactating.
15. Underwent major surgery within 14 days prior to the first dose of ponatinib.
16. Have ongoing or active infection (including known history of human immunodeficiency virus [HIV], hepatitis B virus [HBV], or hepatitis C virus [HCV]).
17. Suffer from any condition or illness that, in the opinion of the Investigator would compromise patient safety or interfere with the evaluation of the safety of the study drug.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Moores UCSD Cancer Center, Site #165, La Jolla, California
  - Southern California Permanente Medical Group, Site #161, San Marcos, California
  - Kaiser Permanente Medical Center, Site #158, Vallejo, California
  - Smilow Cancer Hospital at Yale New Haven, Site #182, New Haven, Connecticut
  - Cancer Institute of Florida, Site #187, Altamonte Springs, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Site #017, Tampa, Florida
  - Emory University, Site # 058, Atlanta, Georgia
  - University of Chicago Medical Center, Site #001, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, Site #138, Indianapolis, Indiana
  - Norton Cancer Institute, Site #142, Louisville, Kentucky
  - University of Maryland, Site #040, Baltimore, Maryland
  - Tufts Medical Center, Site #141, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Site 008, Boston, Massachusetts
  - University of Massachusetts Worcester, Site #152, Worcester, Massachusetts
  - University of Michigan Health System, Site #011, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Site #034, Detroit, Michigan
  - Mayo Clinic, Site #044, Rochester, Minnesota
  - Freeman Cancer Institute, Site #190, Joplin, Missouri
  - Washington University School of Medicine, Site 007, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Site 128, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Site #029, Buffalo, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, Site #006, New York, New York
  - University of Rochester, Site 137, Rochester, New York
  - Duke University Medical Center, Site 003, Durham, North Carolina
  - Jewish Hospital, Site #175, Cincinnati, Ohio
  - Oregon Health & Science University (OHSU), Site 048, Portland, Oregon
  - Hospital of the University of Pennsylvania, Site #013, Philadelphia, Pennsylvania
  - Jeanes Hospital of TUHS, Site #127, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Site #148, Charleston, South Carolina
  - Tennesse Oncology, PLLC, Site # 076, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Site #005, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Site #043, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Site #100, Seattle, Washington